CLINICAL TRIAL: NCT01761461
Title: Phase III Randomized Trial of Adjuvant Chemotherapy With S-1 vs S-1/Oxaliplatin ± Radiotherapy for Completely Resected Gastric Adenocarcinoma : The ARTIST II Trial
Acronym: ARTIST-II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2012-06-061
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — titanium silicide; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): S-1 40-60mg BID (4weeks - 2weeks off) x 8 cycles
  Interventions: Drug: TS-1, oxaliplatin
- Arm B (Active Comparator): {S-1 40-60mg BID (2weeks - 1week off) + Oxaliplatin 130mg/m2 q 3 week} x 8 cycles
  Interventions: Drug: TS-1, oxaliplatin
- Arm C (Active Comparator): {S-1 40-60mg BID (2weeks - 1week off) + Oxaliplatin 130mg/m2 q 3 weeks} x 2 cycles → S-1 40mg BID (2weeks - 1week off - 2weeks)+ RT 45 Gy (5weeks) → Rest for 4 weeks → {S-1 40-60mg BID (2weeks - 1week off) + Oxaliplatin 130mg/m2 q 3 weeks} x 4 cycles
  Interventions: Drug: TS-1, oxaliplatin

INTERVENTIONS:
Drug: TS-1, oxaliplatin

SUMMARY:
The optimal regimen for adjuvant treatment has not been established in GC yet. We plan to compare TS-1, TS-1/oxaliplatin with or without RT in D2 resected gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven gastric or gastroesophageal adenocarcinoma
2. ≥ D2 lymph node dissection, curative gastrectomy
3. Stage II, III (AJCC 2010) with any N (any stage with N0 will be excluded)
4. Age > 19
5. ECOG 0-2
6. No distant metastasis
7. Adequate bone marrow functions (ANC ≥ 1,500/ul, blood platelet ≥ 100,000/ul, haemoglobin ≥ 10g/dl, transfusion allowed)
8. Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
9. liver functions (serum bilirubin ≤ 1.5mg/dl, AST/ALT ≤ 3 times(normal value)
10. Written informed consent
11. Possible oral intake (food, drug)

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study

  1. Active infection requiring antibiotics
  2. Pregnant, lactating women
  3. Concurrent systemic illness not appropriate for chemotherapy
  4. Resection margin (+) at permanent pathology
  5. Pathologic stage I or IV (Ia or Ib according to AJCC 2010)
  6. Inadequate surgery including D0, D1 resection, dissected LNs less than 12
  7. Paraaortic lymph node (+), pathologically proven
  8. women of potential childbearing not employing adequate contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is disease-free survival (DFS). | 3-year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea